CLINICAL TRIAL: NCT04925843
Title: Association Between Fibrinogen Concentration and Intraoperative Bleeding in Liver Transplantation: a Retrospective Observational Study
Brief Title: Fibrinogen and Intraoperative Bleeding in Liver Transplant
Acronym: FIB_TOF
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 19.115
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: End Stage Liver DIsease; Liver Transplant; Complications
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing liver transplant for end-stage liver disease: The investigators propose to conduct a retrospective cohort study to explore the association between fibrinogen concentration and intraoperative bleeding in patients who underwent a liver transplant between July 2008 and January 2021.

SUMMARY:
Liver transplantation is the only treatment for end-stage liver disease. It is a high-risk surgery that can cause heavy intraoperative bleeding. Bleeding and transfusions of blood products are themselves associated with several postoperative complications. Few data have suggested beneficial interventions that can decrease this bleeding. Such interventions are necessary in order to improve these patients' outcomes. In order to better understand the potential therapeutic targets, a better comprehension of the variables associated with such bleeding is essential. Several previous studies have demonstrated a weak association between usual clotting times and bleeding in this population. However, few studies have evaluated the association between the concentration of fibrinogen and bleeding in this population.

The primary objective of this study is to assess the association between preoperative serum fibrinogen concentration and the volume of intraoperative bleeding. The secondary objective is to assess the association between preoperative serum fibrinogen concentration and the number of red blood cell units transfused during the intraoperative and immediate postoperative periods.

The hypothesis of the study is that a low concentration of preoperative fibrinogen will be associated with an increase in intraoperative bleeding and red blood cell transfusions.

DETAILED DESCRIPTION:
All patients who received a liver transplant between July 2008 and January 2021 at the Centre Hospitalier de l'Université de Montréal (CHUM) will be included. The effect of fibrinogen concentration, intraoperative bleeding, intraoperative and postoperative transfusions, as well as postoperative bleeding-related complications and mortality up to 1 year will be assessed. The analysis will be adjusted for several confounding factors, including other coagulation parameters. The main association model will be a multivariable linear regression.

This study will be used to further explore the association between fibrinogen concentration and bleeding in liver transplantation. These results may help certain clinical decisions, without suggesting any potential effect of fibrinogen correction on clinical outcomes. If an association is found, the bases will be put in place to build a clinical trial evaluating the effects of a preemptive transfusion of blood products correcting this value on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing liver transplant.

Exclusion Criteria:

* Use of cryoprecipitate or fresh frozen plasma after measurement of serum fibrinogen concentration prior to arrival in the operating room.
* Amyloid neuropathy or liver cancer
* Fulminant hepatitis
* Retransplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent a liver transplant for a chronic liver disease during the reference period.
Sampling Method: Non-Probability Sample
Enrollment: 612 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss per mass of red blood cells lost | Up to 48 hours after surgery
  In milliliters

SECONDARY OUTCOMES:
Number of red blood cell transfusions during liver transplantation | At the end of surgery
  Count
Number of perioperative red blood cell transfusions | From the beginning of surgery until 48 hours after surgery
  Count
Occurrence of bleeding complications leading to reintervention and / or angioembolization | 30 days after surgery
  Dichotomous
Occurrence of early retransplantation | 30 days after surgery
  Dichotomous
One year survival | One year after surgery
  Time to event

CONTACTS AND LOCATIONS:
Overall Officials: François Martin Carrier, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Carrier FM, Deshetres A, Ferreira Guerra S, Rioux-Masse B, Zaouter C, Lee N, Amzallag E, Joosten A, Massicotte L, Chasse M. Preoperative Fibrinogen Level and Bleeding in Liver Transplantation for End-stage Liver Disease: A Cohort Study. Transplantation. 2023 Mar 1;107(3):693-702. doi: 10.1097/TP.0000000000004333. Epub 2022 Sep 23. PMID 36150121